CLINICAL TRIAL: NCT02657083
Title: Prevention of Hypoglycemia After Exercise Using DreaMed Substance Administration Device in Children and Adolescents With Type 1 Diabetes (The PHYSI-DREAM Study)
Brief Title: Prevention of Hypoglycemia After Exercise Using Closed Loop System in Children and Adolescents With Type 1 Diabetes
Acronym: PHYSI-DREAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ljubljana, Faculty of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PD-MC-01
Record Dates: First submitted 2016-01-12; First posted 2016-01-15 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2016-08

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glucose control using DreaMed MD-AID (Experimental): In this group the subjects use a closed loop system (DreaMed Substance Administration Device) that combines glucose monitoring system (S.C wired sensor, named Sof® Sensor™ or Enlite® Sensor™), which provides real-time interstitial glucose values, with a modern insulin pump (MiniMed® Paradigm® Veo™, Medtronic) and computer algorithm, which directs insulin delivery in response to glucose sensor data.
  Interventions: Device: DreaMed Substance Administration Device
- Glucose control using SAP (Active Comparator): In this group the subjects use a standard treatment (Sensor Augmented Pump), characterised by glucose monitoring system (S.C wired sensor, named Sof® Sensor™ or Enlite® Sensor™) which provides real-time interstitial glucose values and a modern insulin pump (MiniMed® Paradigm® Veo™, Medtronic) without computer algorithm decisions.
  Interventions: Device: Sensor Augmented Pump (SAP)

INTERVENTIONS:
Device: DreaMed Substance Administration Device — 2 exercise days under DreaMed MD-AID control with afternoon exercise (in the time between 16:30 and 19:30).
  New infusion set and two continuous glucose sensors (one for back-up) will be inserted in the subcutaneous tissue of the arm and then calibrated the day before each visit from 3 to 6.
  The continuous glucose sensor continuously will measure interstitial glucose levels and these values will be sent by the Minilink™ via wireless, low-powered, radio frequency to the Paradigm Veo every 5 minutes for up to 6 days.
  The DreaMed MD-AID uses a vendor-supplied and self-developed (communication module) communication application programming interface (API) in order to retrieve glucose / insulin data from the Paradigm Veo and set insulin treatment according to the algorithm decision.
  Arms: Glucose control using DreaMed MD-AID
Device: Sensor Augmented Pump (SAP) — 2 exercise days under Sensor Augmented Pump with afternoon exercise (in the time between 16:30 and 19:30).
  New infusion set and two continuous glucose sensors (one for back-up) will be inserted in the subcutaneous tissue of the arm and then calibrated the day before each visit from 3 to 6.
  The continuous glucose sensor continuously will measure interstitial glucose levels and these values will be sent by the Minilink™ via wireless, low-powered, radio frequency to the Paradigm Veo every 5 minutes for up to 6 days.
  During the exercise the group will turn off the insulin pump and lower their basal insulin for 20% for the next 4 hours after the exercise
  Arms: Glucose control using SAP

SUMMARY:
The Study will compare treatment with Closed Loop (CL) system - DreaMed MD-AID to the standard treatment without computer algorithm decisions - SAP therapy in 20 children and adolescents with Type 1 Diabetes (T1D) during and after afternoon physical activity.

The aims of the study are:

* to demonstrate that the use of DreaMed MD-AID is safe during physical activity
* to investigate the risk of hypoglycemia among children and adolescents with T1D after afternoon exercise during closed-loop control.

DETAILED DESCRIPTION:
This is investigator initiated, single-center, open-label, crossover, randomized, interventional, in-hospital pediatric study, performed at the University Children's Hospital, University Medical Center Ljubljana.

Study duration will be about 4 weeks per subject, 6 month overall. The study will compare Continuous Glucose Monitoring (CGM) based time in hypoglycemia in an intervention arm (Glucose control using DreaMed MD-AID) to a control arm (Glucose control using SAP).

Each arm includes two exercise days with 1 week in-between. Subjects will be randomly assigned to participate first in the intervention arm (10 subjects) or first in the control arm (10 subjects). At the end of the first period patients will be asked to participate in another, i.e. the other arm with at least one week between arms.

Subjects will be instructed to consume a similar diet and avoid caffeine, alcohol, and physical activity in the 48 hours before the exercise day visit.

The start of the run-in period can be scheduled as a separate visit, but not more than 2 days after screening.

All subjects will attend the clinic on six occasions:

* Visit 1: Screening and sensor/pump education, detailed physical examination will be performed, all subject will have to meet inclusion/exclusion criteria.
* Visit 2: Baseline assessment of the DreaMed MD-AID profile, subjects will perform resting electrocardiography (ECG) and determination of the maximal oxygen consumption rate (VO2max) on a cycle ergometer Ganshorn LF8.5G™ and Schiller software, with BG measurements before, at the end of the exercise and 2 hours after exercise. Subjects will be instructed to refrain from physical activity for 48 hours prior to visits 3 - 6.
* Visit 3: 24 hours DreaMed MD-AID or SAP with afternoon exercise (in the time between 16:30 and 19:30): an i.v. catheter will be inserted in the antecubital or cephalic vein (for plasma BG and emergency). Cycle ergometer will be adjusted for each subject (work rate, seat height,..), they will be instructed to pedal at steady rate of 50-60 rotations per minute (RPM).The subjects will cycle for 40 minutes at 55% Vo2max load (starting work rate set to 30 watts (W) with linear loading to reach 55% VO2max on 5:00 minute exercise time) - the aim of this session is to induce delayed hypoglycemia.
* Visit 4: 24 hours DreaMed MD-AID or SAP with afternoon exercise (in the time between 16:30 and 19:30): an i.v. catheter will be inserted in the antecubital or cephalic vein (for plasma BG and emergency). Cycle ergometer will be adjusted for each subject (work rate, seat height,..), they will be instructed to pedal at steady rate of 50-60 rotations per minute (RPM). The subjects will cycle for 40minutes - high intensity interval training (2 - 6 sprints of 20 seconds at 80% VO2max with interval of 6 minutes low-moderate activity (55% VO2max (total of ~40 minutes) between the sprint. The aim of this session is to imitate children's physical activity (bursts of intensive physical activity interspersed with varying intervals of activity of low and moderate intensity.
* Visit 5&6: Same as visits 3 and 4, cross over from DreaMed MD-AID to SAP or vice versa.

During the exercise, a continuous ECG will be recorded and inhaled O2 and exhaled Carbon Dioxide (CO2) will be measured.

BG and lactate will be taken during the exercise visits: at the beginning of the exercise, after every 15 min exercise session, and every half an hour for the next 2 hours thereafter.

All hypoglycemia will be confirmed with SBGM: glucose values <3.3 (60 mg/dl) mmol/l if symptomatic, and all hypoglycemia with self blood glucose monitoring (SBGM) values <2.8 mmol/l (50 mg/dl) (regardless of symptoms) will be treated with rescue carbohydrates as per standard in-hospital procedure (15 g sugar per 10 kg of body weight (BW), re-evaluate and repeat if necessary in 15-30 minutes).

New infusion set and two continuous glucose sensors (one for back-up) will be inserted in the subcutaneous tissue of the arm and then calibrated the day before each visit from 3 to 6.

Schedule for all exercise days will be similar:

* 12:00 hospital admission
* 13:00 lunch
* 13:30 to 16:00 rest
* 16:00 afternoon snack
* 16:30 to 19:30 exercise protocol
* 19:45 dinner
* 21:00 to 7:30 next day: bed time
* 8:00 breakfast.
* 13:00 lunch and end of study

Subjects will have standardized and similar meals on all exercise days (lunch at 13:00, afternoon snack at 16:00, dinner at 19:45, and breakfast at 8:00 the next day), based on the weight, with calculated carbohydrates and calories: 1 gram of carbohydrates per kilogram, the content of the meal according to the recommendation: comprising of 50% carbohydrate, 20% protein, and 30% fat, of which no more than 10% will be saturated fat. During the exercise the SAP group will turn off the insulin pump and lower their basal insulin for 20% for the next 4 hours after the exercise.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed by a parent/legal guardian and informed assent signed by the study participant prior study entry.
* Diagnosed with T1D, as defined by the American Diabetes Association and World Health Organization (ADA/WHO) for at least 1 year prior to study enrolment.
* Documented evidence should exist within the patient history of T1D.
* Age between 10 and 17 years (inclusive) at the time of enrolment.
* Treatment with insulin pump therapy for at least 3 months.
* HbA1C value ≤ 9% based on analysis from the local laboratory at the time of enrolment (A1C testing must follow National Glycohemoglobin Standardization Program (NGSP) standards).
* Willing to follow all study instructions (child and parent should be evaluated as one)
* Availability for the entire study duration and follow-up visits
* Willing to perform daily self-monitoring of blood glucose (SMBG) and required sensor calibrations
* If also present celiac/Hashimoto disease, the disease has to be adequately treated as determined by the investigator
* BMI above 5th centile and below 95th centile for age, respectively.

Exclusion Criteria:

* Concomitant diseases that influence metabolic control (e.g. anemia, significantly impaired hepatic function, renal failure, history of adrenal insufficiency) or other medical conditions, which in the investigator's opinion, may compromise patient safety; Note: Adequately treated thyroid disease and celiac disease do not exclude subjects from enrollment.
* Significant co-morbidity that, in the opinion of the investigators would preclude participation in the study (e.g. current treatment for cancer, mental disorder)
* Any concomitant oral or parenteral glucocorticoids therapy within 1 month prior to screening, or planning to take oral or parenteral glucocorticoids during the study. (Exceptions: Short term oral glucocorticoids up to 7 days, inhaled steroids).
* Any concomitant therapy with antidiabetic agents or other medications, which could be a contraindication to participation in the study by the judgment of the investigator.
* Participation in another study of a medical device or drug that could affect glucose measurements or glucose management or Receipt of any investigational medical product within 1 month prior to screening (Visit 1).
* Female subject of child-bearing potential who is pregnant, breast-feeding, or planning to become pregnant during the study.
* Subject that has known hypoglycemic unawareness or recurrent severe hypoglycemic events with seizure and/or coma (more than two episodes) within 6 months prior to screening.
* History of one or more episodes of Diabetic Ketoacidosis (DKA) requiring hospitalization within a month prior to the screening.
* Current or recent history of alcohol or drug abuse.
* Visual impairment or hearing loss, which in the investigator's opinion, may compromise patient ability to perform study procedures safely (child and parent should be evaluated as a unit).

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
to evaluate the safety and efficacy of blood glucose control using the DreaMed MD-AID in children and adolescents with T1D during and after planned physical activity, in a controlled in-hospital environment. | After all patients completed their 30 days of study treatment.
  Primary endpoint is significant between-group difference (intervention DreaMed MD-AID versus control SAP) in time of hypoglycemia below 3.3 mmol/l (60 mg/dl) during the afternoon exercise and the afternoon/night after (till 13:00 next day) based on sensor glucose readings with a minimum duration of 20 minutes.

SECONDARY OUTCOMES:
to evaluate the physiologic responses and risk of hypoglycemia among children and adolescents with T1D after afternoon exercise during closed-loop control in a controlled in-hospital environment | After all patients completed their 30 days of study treatment.
  * Time of hypoglycemia below 3.9 mmol/l (70 mg/dl) based on sensor glucose readings.
  * Time of hyperglycemia above 13.9 mmol/l (250 mg/dl) based on sensor glucose readings.
  * Time of glucose values within 3.9 - 10 mmol/l (70-180 mg/dl).

CONTACTS AND LOCATIONS:
Overall Officials: Tadej Battelino, Prof, MD, Principal Investigator — University of Ljubljana, Faculty of Medicine
Locations (1):
- University of Ljubljana, Faculty of Medicine, Ljubljana, Slovenia

REFERENCES:
- [Background] American Diabetes Association. Executive summary: Standards of medical care in diabetes--2014. Diabetes Care. 2014 Jan;37 Suppl 1:S5-13. doi: 10.2337/dc14-S005. No abstract available. PMID 24357214
- [Background] Adolfsson P, Nilsson S, Albertsson-Wikland K, Lindblad B. Hormonal response during physical exercise of different intensities in adolescents with type 1 diabetes and healthy controls. Pediatr Diabetes. 2012 Dec;13(8):587-96. doi: 10.1111/j.1399-5448.2012.00889.x. PMID 23173876
- [Background] Beraki A, Magnuson A, Sarnblad S, Aman J, Samuelsson U. Increase in physical activity is associated with lower HbA1c levels in children and adolescents with type 1 diabetes: results from a cross-sectional study based on the Swedish pediatric diabetes quality registry (SWEDIABKIDS). Diabetes Res Clin Pract. 2014 Jul;105(1):119-25. doi: 10.1016/j.diabres.2014.01.029. Epub 2014 Feb 23. PMID 24846445
- [Background] Tsalikian E, Mauras N, Beck RW, Tamborlane WV, Janz KF, Chase HP, Wysocki T, Weinzimer SA, Buckingham BA, Kollman C, Xing D, Ruedy KJ; Diabetes Research In Children Network Direcnet Study Group. Impact of exercise on overnight glycemic control in children with type 1 diabetes mellitus. J Pediatr. 2005 Oct;147(4):528-34. doi: 10.1016/j.jpeds.2005.04.065. PMID 16227041
- [Background] Rosenbauer J, Dost A, Karges B, Hungele A, Stahl A, Bachle C, Gerstl EM, Kastendieck C, Hofer SE, Holl RW; DPV Initiative and the German BMBF Competence Network Diabetes Mellitus. Improved metabolic control in children and adolescents with type 1 diabetes: a trend analysis using prospective multicenter data from Germany and Austria. Diabetes Care. 2012 Jan;35(1):80-6. doi: 10.2337/dc11-0993. Epub 2011 Nov 10. PMID 22074726
- [Background] Hovorka R, Allen JM, Elleri D, Chassin LJ, Harris J, Xing D, Kollman C, Hovorka T, Larsen AM, Nodale M, De Palma A, Wilinska ME, Acerini CL, Dunger DB. Manual closed-loop insulin delivery in children and adolescents with type 1 diabetes: a phase 2 randomised crossover trial. Lancet. 2010 Feb 27;375(9716):743-51. doi: 10.1016/S0140-6736(09)61998-X. Epub 2010 Feb 4. PMID 20138357
- [Background] Ly TT, Breton MD, Keith-Hynes P, De Salvo D, Clinton P, Benassi K, Mize B, Chernavvsky D, Place J, Wilson DM, Kovatchev BP, Buckingham BA. Overnight glucose control with an automated, unified safety system in children and adolescents with type 1 diabetes at diabetes camp. Diabetes Care. 2014 Aug;37(8):2310-6. doi: 10.2337/dc14-0147. Epub 2014 May 30. PMID 24879841
- [Background] Sherr JL, Cengiz E, Palerm CC, Clark B, Kurtz N, Roy A, Carria L, Cantwell M, Tamborlane WV, Weinzimer SA. Reduced hypoglycemia and increased time in target using closed-loop insulin delivery during nights with or without antecedent afternoon exercise in type 1 diabetes. Diabetes Care. 2013 Oct;36(10):2909-14. doi: 10.2337/dc13-0010. Epub 2013 Jun 11. PMID 23757427
- [Background] Phillip M, Battelino T, Atlas E, Kordonouri O, Bratina N, Miller S, Biester T, Stefanija MA, Muller I, Nimri R, Danne T. Nocturnal glucose control with an artificial pancreas at a diabetes camp. N Engl J Med. 2013 Feb 28;368(9):824-33. doi: 10.1056/NEJMoa1206881. PMID 23445093
- [Background] Oron T, Farfel A, Muller I, Miller S, Atlas E, Nimri R, Phillip M. A remote monitoring system for artificial pancreas support is safe, reliable, and user friendly. Diabetes Technol Ther. 2014 Nov;16(11):699-705. doi: 10.1089/dia.2014.0090. Epub 2014 Sep 11. PMID 25211216
- [Background] Dauber A, Corcia L, Safer J, Agus MS, Einis S, Steil GM. Closed-loop insulin therapy improves glycemic control in children aged <7 years: a randomized controlled trial. Diabetes Care. 2013 Feb;36(2):222-7. doi: 10.2337/dc12-1079. Epub 2012 Oct 1. PMID 23033237
- [Background] Elleri D, Allen JM, Kumareswaran K, Leelarathna L, Nodale M, Caldwell K, Cheng P, Kollman C, Haidar A, Murphy HR, Wilinska ME, Acerini CL, Dunger DB, Hovorka R. Closed-loop basal insulin delivery over 36 hours in adolescents with type 1 diabetes: randomized clinical trial. Diabetes Care. 2013 Apr;36(4):838-44. doi: 10.2337/dc12-0816. Epub 2012 Nov 27. PMID 23193217
- [Background] Nimri R, Danne T, Kordonouri O, Atlas E, Bratina N, Biester T, Avbelj M, Miller S, Muller I, Phillip M, Battelino T. The "Glucositter" overnight automated closed loop system for type 1 diabetes: a randomized crossover trial. Pediatr Diabetes. 2013 May;14(3):159-67. doi: 10.1111/pedi.12025. Epub 2013 Feb 28. PMID 23448393
- [Background] Nimri R, Muller I, Atlas E, Miller S, Fogel A, Bratina N, Kordonouri O, Battelino T, Danne T, Phillip M. MD-Logic overnight control for 6 weeks of home use in patients with type 1 diabetes: randomized crossover trial. Diabetes Care. 2014 Nov;37(11):3025-32. doi: 10.2337/dc14-0835. Epub 2014 Jul 30. PMID 25078901
- [Background] Bailey RC, Olson J, Pepper SL, Porszasz J, Barstow TJ, Cooper DM. The level and tempo of children's physical activities: an observational study. Med Sci Sports Exerc. 1995 Jul;27(7):1033-41. doi: 10.1249/00005768-199507000-00012. PMID 7564970
- [Background] Guelfi KJ, Jones TW, Fournier PA. The decline in blood glucose levels is less with intermittent high-intensity compared with moderate exercise in individuals with type 1 diabetes. Diabetes Care. 2005 Jun;28(6):1289-94. doi: 10.2337/diacare.28.6.1289. PMID 15920041
- [Background] Bussau VA, Ferreira LD, Jones TW, Fournier PA. A 10-s sprint performed prior to moderate-intensity exercise prevents early post-exercise fall in glycaemia in individuals with type 1 diabetes. Diabetologia. 2007 Sep;50(9):1815-1818. doi: 10.1007/s00125-007-0727-8. Epub 2007 Jun 22. PMID 17583795
- [Background] Bussau VA, Ferreira LD, Jones TW, Fournier PA. The 10-s maximal sprint: a novel approach to counter an exercise-mediated fall in glycemia in individuals with type 1 diabetes. Diabetes Care. 2006 Mar;29(3):601-6. doi: 10.2337/diacare.29.03.06.dc05-1764. PMID 16505513
- [Background] Tonoli C, Heyman E, Roelands B, Buyse L, Cheung SS, Berthoin S, Meeusen R. Effects of different types of acute and chronic (training) exercise on glycaemic control in type 1 diabetes mellitus: a meta-analysis. Sports Med. 2012 Dec 1;42(12):1059-80. doi: 10.1007/BF03262312. PMID 23134339
- [Background] Robertson K, Riddell MC, Guinhouya BC, Adolfsson P, Hanas R; International Society for Pediatric and Adolescent Diabetes. ISPAD Clinical Practice Consensus Guidelines 2014. Exercise in children and adolescents with diabetes. Pediatr Diabetes. 2014 Sep;15 Suppl 20:203-23. doi: 10.1111/pedi.12176. No abstract available. PMID 25182315
- [Background] Pivovarov JA, Taplin CE, Riddell MC. Current perspectives on physical activity and exercise for youth with diabetes. Pediatr Diabetes. 2015 Jun;16(4):242-55. doi: 10.1111/pedi.12272. Epub 2015 Mar 9. PMID 25754326
- [Derived] Dovc K, Macedoni M, Bratina N, Lepej D, Nimri R, Atlas E, Muller I, Kordonouri O, Biester T, Danne T, Phillip M, Battelino T. Closed-loop glucose control in young people with type 1 diabetes during and after unannounced physical activity: a randomised controlled crossover trial. Diabetologia. 2017 Nov;60(11):2157-2167. doi: 10.1007/s00125-017-4395-z. Epub 2017 Aug 24. PMID 28840263